CLINICAL TRIAL: NCT05104931
Title: A Phase 1, Single-Centre, Part-Crossover, OpenLabel, Partially-Randomised Study Designed to Evaluate the PK Profile of Piroxicam Following Administration of Nanoformed Oral IR Piroxicam Tablet and an IR Reference Product in Healthy Subjects
Brief Title: PK Evaluation of a Nanoformed Oral IR Piroxicam Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanoform Finland Plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNICORN
Record Dates: First submitted 2021-03-28; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Piroxicam; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nanoformed Piroxicam IR Tablet (Experimental): orally delivered nanoformed piroxicam immediate release tablets (20mg)
  Interventions: Drug: Nanoformed Piroxicam IR Tablet
- Felden (piroxicam) Tablets (Active Comparator): orally delivered Felden (piroxicam) tablets (20mg)
  Interventions: Drug: Felden (piroxicam) Tablets
- Brexidol (piroxicam) Tablets (Active Comparator): orally delivered Brexidol (piroxicam) tablets (20mg)
  Interventions: Drug: Nanoformed Piroxicam IR Tablet; Drug: Brexidol (piroxicam) Tablets

INTERVENTIONS:
Drug: Nanoformed Piroxicam IR Tablet — Orally delivered Nanoformed Piroxicam
  Other Names: Orally delivered Nanoformed Piroxicam IR tablet
  Arms: Brexidol (piroxicam) Tablets; Nanoformed Piroxicam IR Tablet
Drug: Felden (piroxicam) Tablets — orally delivered Felden (reference) tablets
  Other Names: orally delivered Felden (piroxicam) tablets
  Arms: Felden (piroxicam) Tablets
Drug: Brexidol (piroxicam) Tablets — orally delivered Brexidol (reference) tablets
  Other Names: orally delivered Brexidol (piroxicam) tablets
  Arms: Brexidol (piroxicam) Tablets

SUMMARY:
Piroxicam is a nonsteroidal anti-inflammatory medication and currently used to treat pain and inflammation caused by osteoarthritis or rheumatoid arthritis. The aim of this study is to study the pharmacokinetic behaviour of the new nanoformed 20mg tablet formulation of piroxicam in comparison with a reference 20mg piroxicam tablet formulation. The target of nanoforming is to improve the pharmacokinetic properties of drugs with low solubility, potentially leading to the use of lower doses with concomitant improvements in safety and tolerability. Piroxicam is an appropriate candidate to demonstrate the benefits of nanoforming due to its physiochemical properties. The efficacy of the Nanoformed Piroxicam is evaluated in comparison to the reference product Felden® Tabs 20 mg. The study also is conducted with a second reference product, Brexidol® 20 mg, or a nanoformed piroxicam tablet of a different strength, or study the effect of food intake on the absorption of the nanofomed piroxicam tablet. The study is conducted with healthy volunteers.

DETAILED DESCRIPTION:
This is a single-centre, open-label, partly-randomised, part-cross-over up to three-period, comparative bioavailability study in healthy male and female subjects, designed to investigate the pharmacokinetic (PK) properties and safety of Nanoformed Piroxicam Immediate Release (IR) Tablet, 5 - 20 mg and Felden® (piroxicam) Tablets 20 mg (reference) with an optional Brexidol® (piroxicam) Tablets 20 mg (alternative reference; optional in Period 3. Subjects will receive single oral doses of the investigational medicinal product across up to 3 treatment periods in either the fasted or fed state (optional in Period 3 only). Subjects will be randomised to 1 of 2 treatment sequences across Periods 1 and 2 which will be dosed in the fasted state. Following completion of Period 2, there will be an interim analysis of the PK and safety data generated from both previous periods to decide whether to proceed to an optional Period 3 and, if progression is made, to dose the Nanoformed Piroxicam IR Tablet, 5 - 20 mg in the fed state, an alternative dose level of Nanoformed Piroxicam IR Tablet, 5 - 20 mg in the fasted state or an alternative reference product in the fasted state in Period 3 (optional). The maximum dose of piroxicam that will be administered in any period of the study is 20 mg. For Period 3, if the Nanoformed Piroxicam IR Tablet, 5 - 20 mg formulation is selected, the dose will be selected from a bracketing dose range of 5 to 20 mg. Each period will follow the same study design. There will be a minimum washout of 12 days between each product administration. It is expected that the study will be executed in a single group, requiring a total of 3 study periods.

The study is exploratory and no formal sample size calculation has been made. Based on experience from previous studies of a similar design, a total of 12 subjects are to be enrolled and a minimum of 8 evaluable subjects are considered sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Aged 18 to 55 years inclusive at the time of signing informed consent
* Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to adhere to the contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
* Subjects who are, or are immediate family members of, a study site or sponsor employee
* Evidence of current SARS-CoV-2 infection
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months. A positive urine cotinine test at screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Females who are pregnant or lactating (all female subjects must have a negative urine pregnancy test)
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* History of clinically significant cardiovascular (including ischaemic heart disease, peripheral arterial disease, heart failure), renal, hepatic, dermatological, chronic respiratory (including asthma) or neurological or psychiatric disorder, as judged by the investigator
* History of gastro-intestinal ulceration, bleeding or perforation
* History of gastrointestinal disorders that predispose to bleeding disorders such as ulcerative colitis, Crohn's disease, gastrointestinal cancers or diverticulitis
* Subjects with active peptic ulcer, inflammatory gastrointestinal disorder or gastrointestinal bleeding
* Subjects with a history of cholecystectomy or gall stones
* History of adverse reactions or allergy associated with any drug
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* History of previous serious allergic drug reaction of any type, especially cutaneous reactions such as erythema multiforme, Stevens-Johnson syndrome, toxic epidermal necrolysis
* Previous skin reaction (regardless of severity) to piroxicam, other NSAIDs and other medications
* Subjects in whom aspirin and other NSAIDs induce the symptoms of asthma, nasal polyps, angioedema or urticaria
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day or hormonal replacement therapy [HRT]/hormonal contraception) in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator
* Concomitant use of other NSAIDs, including cyclooxygenase-2 inhibitors, selective NSAIDs and acetylsalicylic acid at analgesic doses
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Plasma Concentration (Cmax) of piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet 5 - 20 mg and Felden (piroxicam) Tablets 20mg (reference) in healthy subjects in the fasted state. | 72 hours
  To determine the pharmacokinetics and relative bioavailability of piroxicam over a 72h period following administration of single oral doses of Nanoformed Piroxicam IR Tablet 5 - 20 mg and Felden (piroxicam) Tablets 20mg (reference) in healthy subjects in the fasted state by determining the Maximum Plasma Concentration (Cmax).
To determine the Area Under the drug Concentration of piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet 5 - 20 mg and Felden (piroxicam) Tablets 20mg (reference) in healthy subjects in the fasted state. | 72 hours
  To determine the pharmacokinetics and relative bioavailability of piroxicam over a 72h period following administration of single oral doses of Nanoformed Piroxicam IR Tablet 5 - 20 mg and Felden (piroxicam) Tablets 20mg (reference) in healthy subjects in the fasted state by determining the Area Under the drug Concentration time curve over 1 hour (AUC(0 1h)), AUC from time 0 to the time of last measurable concentration (AUC(0 last)) and AUC from time 0 extrapolated to infinity (AUC(0-inf)).
To determine the time to Cmax (Tmax) of piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet 5 - 20 mg and Felden (piroxicam) Tablets 20mg (reference) in healthy subjects in the fasted state. | 72 hours
  To determine the pharmacokinetics and relative bioavailability of piroxicam over a 72h period following administration of single oral doses of Nanoformed Piroxicam IR Tablet 5 - 20 mg and Felden (piroxicam) Tablets 20mg (reference) in healthy subjects in the fasted state by determining the time to Cmax (Tmax).

SECONDARY OUTCOMES:
Number of participants that report adverse events (AEs) coded using MedDRA v23.1, pre-dose and 48-72h post-dose, for determining safety and tolerability. | 72 hours
  To assess additional safety and tolerability information for piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet, 5 - 20mg in healthy subjects by assessing and reporting adverse events (AEs)
To assess additional safety and tolerability information for piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet, 5 - 20mg in healthy subjects by assessing and reporting supine electrocardiograms | 72 hours
  To assess and report 12 lead supine electrocardiogram-measured P-wave pre-dose and 48-72h post-dose, for determining safety and tolerability.
To assess additional safety and tolerability information for piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet, 5 - 20mg in healthy subjects by assessing and reporting supine electrocardiograms | 72 hours
  To assess and report 12 lead supine electrocardiogram-measured QT Interval pre-dose and 48-72h post-dose, for determining safety and tolerability.
To assess additional safety and tolerability information for piroxicam following administration of single oral doses of Nanoformed Piroxicam IR Tablet, 5 - 20mg in healthy subjects by assessing and reporting supine electrocardiograms | 72 hours
  To assess and report 12 lead supine electrocardiogram-measured QRS Complex pre-dose and 48-72h post-dose, for determining safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Evans, MBChB, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom